CLINICAL TRIAL: NCT00172900
Title: MR Spectroscopy and Diffusion Tensor Imaging of White Matter in Alzheimer's Disease
Brief Title: MRS and DTI of White Matter in Alzheimer's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700320
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-12-21 (Estimated); Status verified 2005-06

CONDITIONS: Alzheimer's Disease; Vascular Dementia
Keywords: Diffusion tensor imaging; MR spectroscopy; dementia; white matter
MeSH Terms: conditions — Alzheimer Disease; Dementia, Vascular; Dementia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The white matter change of the Alzheimer's disease could be studied by diffusion tensor image and MR spectroscopy to see the microstructral and biochemical change.

ELIGIBILITY:
Inclusion Criteria:

* probable Alzheimer's disease or subcortica type vascular dementia

Exclusion Criteria:

* large vessel infarct, major trauma

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Fang Chen, MD, Study Director — Department of Medical Imaging, National Taiwan University Hospital
Locations (1):
- Department of Medical Imaging, National Taiwan University Hospital, Taipei, Taiwan